CLINICAL TRIAL: NCT00433407
Title: A Study to Assess HER2-Specific T Cell Responses in Patients Receiving Trastuzumab for Solid Tumor Treatment
Brief Title: T-Cell Response in Patients Receiving Trastuzumab and/or Chemotherapy for HER2-Positive Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449959; UCLA-0505075-01
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer; recurrent breast cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Sarcoma; Breast Neoplasms, Male; Carcinoma, Ovarian Epithelial; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trastuzumab (Experimental): blood sample collected on different days from patients receiving trastuzumab
  Interventions: Biological: trastuzumab

INTERVENTIONS:
Biological: trastuzumab

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment. It may also help the study of cancer in the future.

PURPOSE: This laboratory study is looking at blood samples from patients receiving trastuzumab and/or chemotherapy for HER2-positive solid tumors to assess T-cell response.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess T-cell activation in blood samples of patients receiving trastuzumab (Herceptin®) and/or chemotherapy for HER2-positive solid tumors.

OUTLINE: Blood samples are collected from patients at baseline and on days 21, 42, and 84 of trastuzumab (Herceptin®)/chemotherapy. Patients may be contacted 3-6 months after completion of trastuzumab/chemotherapy to donate another blood specimen.

Blood samples are examined for T-cell proliferation and intracellular cytokine production. CD8 T-cell response, HER2/neu-specific antibody titers, and skin hypersensitivity test responses are also measured.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid epithelial tumor, including, but not limited to, the following:

  * Breast cancer
  * Ovarian cancer
  * Lung cancer
  * Uterine cancer
  * Prostate cancer
* HER2/neu-positive disease by immunohistochemistry or fluorescent in situ hybridization
* Must be receiving trastuzumab (Herceptin®) and/or chemotherapy (e.g., paclitaxel, docetaxel, fluorouracil, or estramustine)

PATIENT CHARACTERISTICS:

* Absolute neutrophil count > 1,000/mm^3
* Absolute lymphocyte count > 400/mm^3
* Platelet count > 90,000/mm^3
* Hemoglobin > 8 g/dL

PRIOR CONCURRENT THERAPY:

* No other chemotherapy within the past 4 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
T-cell activation in blood samples | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States